CLINICAL TRIAL: NCT02778776
Title: Effect of Administration of Combination Metformine/Inulin Versus Metformine on Patients With Prostate Benign Hyperplasia and Metabolic Syndrome Syndrome
Brief Title: Combination of Metformine/Inulin Versus Metformin on Prostate Benign Hyperplasia in Metabolic Syndrome
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Centro Universitario de Ciencias de la Salud, Mexico (Other)
Responsible Party: Principal Investigator, Fernando Grover Paez, Fernando Grover-Paez, PhD, Centro Universitario de Ciencias de la Salud, Mexico
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CUCS-INTEC-MV-HBP-001
Record Dates: First submitted 2016-05-18; First posted 2016-05-20 (Estimated); Last update posted 2016-05-20 (Estimated); Status verified 2016-05

CONDITIONS: Metabolic Syndrome
Keywords: Metformin; Agave Inulin; METS; Inflammation parameters; Urodynamic parameters; Prostate hyperplasia
MeSH Terms: conditions — Metabolic Syndrome; Prostatic Hyperplasia | interventions — Metformin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Agave inulin + Metfomin (Experimental): 5 g of Agave inulin powder every 12 hrs + 500 mg tablet of metformin every 24 hrs
  Interventions: Drug: Metformin; Dietary Supplement: Agave inulin
- Metformin + Placebo of agave inulin (Active Comparator): 500 mg tablet of metformin every 24 hrs + 5 g every 12 hrs of calcinated magnesia powder
  Interventions: Drug: Metformin; Other: Placebo of agave inulin
- Agave Inulin+Placebo of Metformin (Active Comparator): 5 g of agave inulin powder every 12 hrs + 500 mg tablet of calcinated magnesia as metformin placebo every 24 hrs
  Interventions: Dietary Supplement: Agave inulin; Other: Metformin placebo
- Placebo of Inulin + Placebo of Metformin (Placebo Comparator): 5 g of calcinated magnesia powder every 12 hrs + 500 mg tablet of calcinated magnesia every 24 hrs
  Interventions: Other: Placebo of agave inulin; Other: Metformin placebo

INTERVENTIONS:
Drug: Metformin — Metfomin in tablet presentation of 500 mg
  Other Names: GLUCOPHAGE
  Arms: Agave inulin + Metfomin; Metformin + Placebo of agave inulin
Dietary Supplement: Agave inulin — Oligofructan in powder obtained from agave plant, it was given to each patient a full 10 mg container.
  Arms: Agave Inulin+Placebo of Metformin; Agave inulin + Metfomin
Other: Placebo of agave inulin — Calcinated magnesia powder
  Arms: Metformin + Placebo of agave inulin; Placebo of Inulin + Placebo of Metformin
Other: Metformin placebo — Calcinated magnesia tablet
  Arms: Agave Inulin+Placebo of Metformin; Placebo of Inulin + Placebo of Metformin

SUMMARY:
Type 2 diabetes mellitus, insulin resistance, visceral obesity and disorders of lipid metabolism, especially triglyceride and hypertension are metabolic disorders that play a central role in pathophysiology of metabolic syndrome, and ultimately, the cardiovascular morbidity and mortality associated with atherosclerosis, such as myocardial infarction, cerebral vascular events, vascular dementia, heart failure and end stage renal disease. Recently other complications related with hyperinsulinemia like the prostate benign hypertrophy (BPH). Metformin is the treatment of choice in patients with metabolic syndrome, given its low cost and comparable pharmacological effects to the tiazolinedionas (eg pioglitazone), decreasing hyperinsulinemia, insulin resistance, concentration of free fatty acids and triglycerides, also it produces moderate weight loss, improving the metabolic profile triglcerides atherogenic lipid and carbohydrate and delaying the onset of diabetes mellitus in individuals with impaired fasting glucose.

A second option for risk reduction would be the addition of inulin fiber type as it has been demonstrated some metabolic effects on benefices lipid metabolism and carbohydrate.

It is expected that combination of metformin with inulin produce a beneficial effect through farmacological synergism and the impact on fisiopatological changes of metabolic syndrome that potentially is considered as an important risk factor for prostate growth.

DETAILED DESCRIPTION:
The main objective is to evaluate the effect of the combination of metformin / inulin on clinical, urodynamic parameters as well as metabolic and inflammatory profile in patients with benign prostate hypertrophy and metabolic syndrome.

The investigators conducted a double-blind trial, randomized, on 4 groups, each group with 15 male and female patients of 40 to 80 years of age with METS diagnosed by IDF criteria and clinical diagnose of HBP. Randomization will determine who will receive the intervention during 12 week trial, each group will be like:

Group (A) intervention with combination metformin/ inulin: 15 individuals recieved combination of metformin/ agave inulin in a dosis of 500 mg / 10 grs per 24hrs during 12 weeks.

Group (B) Metformin plus Placebo of agave inulin: 15 individuals recieved Metformin in a dosis of 500mg per day (with the first bite of the second meal) plus homologue placebo of agave inulin (calcinated magnesia) in a dosis of 10grs each 24 hrs during 12 weeks.

Group (C) agave inulin plus placebo of Metformin: 15 indivuduals recieved agave inulin in a dosis of 10grs per 24hrs plus homologate placebo of metformin (calcinated magnesia) in a dosis of 500 mg per day (with the first bite of the second meal) during 12 weeks.

Group (D) Placebo of agave inulin plus Placebo of Metformin: homologate placebo of agave inulin (calcinated magnesia) in a dosis of 10 grs each 24 hrs plus homologate placebo of metformin (calcinated magnesia capsules) in a dosis of 500 mg per day (with the first bite of the second meal) during 12 weeks.

The clinical findings and laboratory test include a metabolic profile and biosafety, will be baseline and at 12 weeks.

Clinical components of Mets like antropometrics parameters, fasting glucose, fasting insulin, blood lipids, clinical finding of HBP and inflammation parameters and adipocitocins, IGF-1, insulin, prostatic specific antigen. Adverse events and adherence to treatment will be documented. Statistical analysis: Mann-Whitney U Test and Wilcoxon exact test. It is considered with significance at p<0.05.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of metabolic syndrome by IDF criteria

  * a person to be defined as having the metabolic syndrome they must have: Central obesity (defined as waist circumference* with ethnicity specific values) ≥80 cm in females and ≥90 cm in males; and plus any two of the following four factors:
  * Raised triglycerides ≥ 150 mg/dL (1.7 mmol/L) or specific treatment for this lipid abnormality Reduced HDL cholesterol
  * < 40 mg/dL (1.03 mmol/L) in males < 50 mg/dL (1.29 mmol/L) in females or specific treatment for this lipid abnormality
  * Raised blood pressure systolic BP ≥ 130 or diastolic BP ≥ 85 mm Hg or treatment of previously diagnosed hypertension
  * Raised fasting plasma glucose (FPG) ≥ 100 mg/dL (5.6 mmol/L), or previously diagnosed type 2 diabetes
* Age ranging from 40 to 80 years old
* Male patients
* Informed written consent

Exclusion Criteria:

* Kidney disease
* Hepatic disease
* Thyroid disease
* Diabetes mellitus
* Ischemic heart disease
* Drug consumption
* Alcohol consumption of more than 2 ounces daily
* Consumption of drugs that intervene with lipid or glucose metabolism 2 months before
* Blood pressure >160/100mmHg.
* Lack of adherence to treatment (adherence <80%)

Ages: 40 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2013-01; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
International Prostate Symptom Score (I-PSS) | 12 weeks
  before and after intervention questionnaire

SECONDARY OUTCOMES:
Change of waist circumference | 12 weeks
  Measured with a non elastic tape at baseline and after intervention
Change of body mass index | 12 weeks
  before and after intervention using a tetrapolar bioelectrical impedance analyzer (body composition analyzer TBF-215 - Tanita)
Change from baseline in Peripheral systolic blood pressure | 12 weeks
  Before and after intervention using a digital sphygmomanometer
Change from baseline in Peripheral diastolic blood pressure | 12 weeks
  Before and after intervention using a digital sphygmomanometer
Change of HOMA-IR from base line to 12 weeks | 12 weeks
  Before and after intervention by using the formula for the homeostasis model assessment β-cell function index: 20 x fasting insulin (µU/Ml)/fasting glucose (mmol/L) - 3.5.
Change from baseline in High-density lipoprotein cholesterol at 12 weeks | 12 weeks
  Before and after intervention by spectrophotometry
Change from Baseline in Triglycerides at 12 weeks | 12 weeks
  Before and after intervention by spectrophotometry
Change from Baseline in Total cholesterol at 12 weeks | 12 weeks
  Before and after intervention by spectrophotometry
Change from Baseline in Fasting plasma glucose at 12 weeks | 12 weeks
  Before and after intervention by glucose oxidase
qmax urine flow rate | 12 weeks
  before and after intervention by uroflowmetry
prostate serum antigen | 12 weeks
  before and after intervention by colorimetry

CONTACTS AND LOCATIONS:
Overall Officials: FERNANDO GROVER, PhD, Principal Investigator — Institute of Experimental and Clinical Therapeutics (INTEC), CUCS, University of Guadalajara
Locations (1):
- Universidad de Guadalajara, Guadalajara, Jalisco, México, Mexico

IPD SHARING:
Plan to Share IPD: No